CLINICAL TRIAL: NCT06381570
Title: VICTORY: A Pilot Study to Investigate Safety and Efficacy of Weekly Combination of Intravenous Vinblastine With Oral Type II RAF Inhibitor Tovorafenib in Pediatric Patients With Recurrent/Progressive RAF Altered Low Grade Gliomas
Brief Title: Pilot Study of Vinblastine and Tovorafenib in Pediatric Patients With Recurrent/Progressive RAF Altered Low Grade Gliomas
Acronym: VICTORY
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Daniel Morgenstern (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Sponsor-Investigator, Daniel Morgenstern, Senior Medical Officer, The Hospital for Sick Children
Organization: The Hospital for Sick Children (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICTORY/OZM-138
Record Dates: First submitted 2024-04-10; First posted 2024-04-24 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Low-grade Glioma
Keywords: RAF altered; non-NF1
MeSH Terms: interventions — tovorafenib; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (single arm study) (Experimental)
  Interventions: Drug: Tovorafenib; Drug: Vinblastine

INTERVENTIONS:
Drug: Tovorafenib — Tovorafenib for oral dosing is provided as an immediate-release tablet in 100 mg strength. The 100 mg tablets are red to yellowish red oval tablets. All products are labeled tovorafenib. In addition, tovorafenib is provided as a powder for reconstitution (PfR) in bottles (430mg per bottle to deliver 300 mg dose). Upon reconstitution with water, the concentration is 25 mg/mL.
  Vinblastine is administered by intravenous route as IV push, sites to follow local administration guidelines, once weekly (central line, but peripheral line is also permitted)
  Other Names: Vinblastine
Drug: Vinblastine — vinblastine in combination with tovorafenib

SUMMARY:
This is a Pilot, multicenter, open-label study of patients less than or equal to 25 years, with recurrent or progressive LGG harboring a CRAF or BRAF alteration, including BRAF V600 mutations and KIAA1549: BRAF fusions. Patients with BRAF or CRAF alterations will be identified through molecular assays as routinely performed at Clinical Laboratory Improvement Amendments (CLIA) of 1988 or other similarly certified laboratories.

The study will be conducted in two sequential phases:

Phase A: A Feasibility (combination dose finding) phase, followed by Phase B: An Efficacy phase. The maximum tolerated dose (MTD)/Recommended Phase 2 Dose (RP2D) of the combination as determined in Phase A would be the dose used in Phase B. The patients on Phase A who were below the MTD/RP2D would be eligible for intra-patient dose escalation to MTD/RP2D subject to criteria outlined later

DETAILED DESCRIPTION:
Phase A (Feasibility Phase) A feasibility phase will be conducted to establish the maximum tolerated dose (MTD/RP2D) of the combination of vinblastine + tovorafenib using the Rolling 6 design.

Patients will receive vinblastine and tovorafenib on Days 1, 8, 15, 22 of each cycle for a total duration of 17 cycles followed by 7 additional cycles of tovorafenib alone. One cycle of protocol therapy is 28 days.

Treatment cycles will repeat every 28 days for a total of 24 cycles in the absence of disease progression or unacceptable toxicity. Patients will undergo radiographic evaluation of their disease at the end of every third cycle, starting with the end of Cycle 3.

The RP2D of tovorafenib of 420 mg/m2 once weekly (not exceeding 600 mg) in combination with vinblastine (4mg/m2) will be used as the starting dose and will be de-escalated/escalated as per Table 4. Dose of tovorafenib will not be escalated further.

Patients will be treated on protocol therapy for a total of 24 cycles, the vinblastine and tovorafenib for a total duration of 17 cycles followed by 7 additional cycles of alone tovorafenib, unless disease progression, unacceptable toxicity occurs, or withdrawal from the study occurs. Missed doses of either vinblastine or tovorafenib will not be made up.

Phase B (Expansion/Efficacy Phase) Once the MTD/RP2D of the combination, vinblastine + tovorafenib has been established, the expansion/efficacy phase will be initiated at the dose determined in Phase A.

Patient will receive vinblastine and tovorafenib weekly on Days 1, 8, 15, 22 of each cycle at dose determined in Phase A for a total duration of 17 cycles followed by 7 additional cycles of tovorafenib alone. One cycle of protocol therapy is 28 days.

Treatment cycles will repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients will undergo radiographic evaluation of their disease at the end of every third cycle, starting with the end of Cycle 3.

Patients will be treated on protocol therapy for a total of 24 cycles, the vinblastine and tovorafenib for a total duration of 17 cycles followed by 7 additional cycles of alone tovorafenib, unless disease progression or unacceptable toxicity occurs, unless disease progression, unacceptable toxicity or withdrawal from study occurs. Missed doses of either vinblastine or tovorafenib will not be made up.

ELIGIBILITY:
Inclusion Criteria:

1. Age

   a) Patients must be less than or equal to 25 years of age at the time of enrollment.
2. Study Group

   a) Progressive/Recurrent LGG (non-NF1) with documented BRAF or CRAF alteration as identified through molecular assays as routinely performed at CLIA or other similar certified laboratories.
3. Diagnosis

   1. All patients must have pathological confirmation of low-grade glioma with BRAF or CRAF alteration.
   2. Patient must have progressive or recurrent LGG.
   3. Must have at least 1 measurable lesion, as defined by RANO-LGG criteria.
   4. Eligible histologies will include all tumors considered low-grade glioma or low-grade astrocytoma (WHO grade I and II) by WHO classification of Tumors of the Central Nervous system -5th edition revised with exception of subependymal giant cell astrocytoma.
4. Prior Therapy

   1. Must have received at least 1 line of systemic therapy prior (at least a vinca alkaloid and/or single agent carboplatin and/or a MEK or BRAF inhibitor) and have documented evidence of radiographic progression.
   2. Patients must have fully recovered from the acute toxic effects (≤ Grade I) of all prior anticancer chemotherapy and have undergone the following washout periods, as applicable.

   i. Myelosuppressive chemotherapy: At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea) ii. Radiation therapy (XRT): Radiation therapy to the measurable lesion(s) must be completed at least 6 months prior to administration of combination therapy. Patients who have documented radiographic progression less than 6 months from radiotherapy in 1 or more measurable lesions are eligible. At least 2 weeks after the last dose fraction of XRT to the non-target lesion.

   iii. Investigational agent or any other anticancer therapy not defined above: At least four weeks prior to planned start of combination therapy, or five half-lives, whichever is shorter.

   iv. Patients must have recovered from acute effects of any prior surgery. v. Chronic toxicities from prior anticancer therapy must be stable as per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 Grade ≤ 2, except ongoing retinopathy which must be ≤ Grade 1.
5. Performance Level

   a) Karnofsky (those 16 years and older) or Lansky (those younger than 16 years) performance score of at least 50. Patients who are unable to walk because of paralysis, but who are able to sit in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
6. Tumor Tissue Sample Confirmation that an archival tumor tissue sample is available. If an archival tumor tissue sample is not available, a fresh biopsy should be performed at baseline. Submission of tumor tissue and a blood sample are mandatory and must be submitted within 14 days from enrollment onto the study and prior to initiation of treatment. Biopsy may be either at initial diagnosis or recurrence.
7. Organ function

   a) Adequate bone marrow function defined as: i. Absolute neutrophil count ≥ 1000/mm3 ii. Platelet count (unsupported) ≥ 100 x 109/L (transfusions allowed per institutional guidelines; last transfusion > 2 weeks prior to enrollment) iii. Hemoglobin (unsupported)≥ 10.0 g/dL (transfusions allowed per institutional guidelines; last transfusion > 4 weeks prior to enrollment) iv. Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (e.g., Neulasta®) or 7 days for short-acting growth factor.

   b) Adequate hepatic and renal function defined as: i. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age (patients with documented Gilbert's disease may be enrolled with sponsor approval and total bilirubin ≤ 2 x ULN) ii. Serum glutamic-pyruvic transaminase (SGPT)/alanine aminotransferase (ALT) ≤ 2.5 x ULN iii. Serum glutamic-oxaloacetic transaminase (SGOT)/aspartate transaminase (AST) ≤ 2.5 x ULN iv. Serum creatinine within normal limits or estimated glomerular filtration rate

   ≥ 60 ml/min/1.73 m2 based on local institutional practice for determination. c) Thyroid functions tests within institutional normal range. Patients on a stable dose of thyroid replacement therapy for a minimum of 3 weeks before starting therapy are eligible.

   d) Adequate cardiac function defined as: i. Left ventricular ejection fraction (LVEF) of ≥ 50% as measured by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan, or fractional shortening (FS) ≥ 25% (Tissot et al., 2018) as measured by ECHO, within 14 days before enrollment (while not receiving medications for cardiac function). If normal practice at the institution is to provide the LVEF result as a range of values, then the upper value of the range will be used to determine the result.

   ii. QTc (by Fridericia's formula) < 470ms as measured by electrocardiogram (ECG) within 14 days before enrollment (while not receiving medications for cardiac function).

   e) Adequate central nervous system (CNS) function defined as: i. Patients with seizures should be stable and not have experienced a significant increase in seizure frequency within 14 days prior to enrollment.

   ii. Patients with neurologic deficits should have deficits that are stable for a minimum of 14 days prior to enrollment.

   iii. Patients receiving steroids for tumor-associated symptoms must be on a stable dose (e.g., no initial/loading dose, no increase or decrease) for 14 days prior to enrollment.
8. Study specific

   1. Baseline ophthalmology assessment within 28 days of study enrollment.
   2. MRI assessment within 28 days of study enrollment. MRI done for clinical indication but within the window for study would be permitted as baseline.
   3. Ability to comply with treatment, laboratory monitoring, and required clinic visits for the duration of study participation.
   4. Willingness of male and female patients with reproductive potential to use double effective birth control methods, defined as one used by the patient and another by his/her partner, for the duration of treatment and for 180 days following the last dose of study drug. Effective birth control methods are described in Appendix H.
   5. Ability to swallow tablets or liquid, or gastric access via a nasal or gastric tube.
   6. Patient is able to start treatment within 14 working days of screening.
   7. Parent/guardian of child or adolescent patient has the ability to understand, agree to, and sign the study ICF and applicable pediatric assent form before initiation of any protocol related procedures; patient has the ability to give assent, as applicable, at the time of parental/guardian consent.

Exclusion Criteria:

* Patients meeting any of the following criteria are to be excluded from study participation:

  1. Patient's tumor has additional previously known activating molecular alterations, other than BRAF or CRAF.
  2. Known or suspected diagnosis of neurofibromatosis Type 1 (NF-1) via genetic testing or current diagnostic clinical criteria.
  3. History of any major disease, other than the diagnosis of LGG, that might interfere with safe protocol participation.
  4. Patient with a history or current evidence of central serous retinopathy (CSR), retinal vein occlusion (RVO), or ophthalmopathy present at baseline who would be considered a risk factor for CSR or RVO. Ophthalmological findings secondary to long-standing optic pathway glioma (such as visual loss, optic nerve pallor, or strabismus) will NOT be considered a significant abnormality for the purposes of this study.
  5. Major surgery within 14 days (2 weeks) prior to enrollment (does not include central venous access, cyst fenestration or cyst drainage, or ventriculoperitoneal shunt placement or revision).
  6. Clinically significant active cardiovascular disease, or history of myocardial infarction, or deep vein thrombosis/pulmonary embolism within 6 months prior to enrollment, ongoing cardiomyopathy, or current prolonged QT interval corrected for heart rate by Fridericia's formula (QTcF) interval > 470 ms based on triplicate ECG average.
  7. Concomitant medications that are strong inhibitors or inducers of CYP2C8 or CYP3A4 within 14 days before initiation of therapy. Concomitant medications that are substrates of BCRP with a narrow therapeutic index within 14 days before initiation of therapy
  8. Current enrollment in any other investigational treatment study. Participation on a concurrent observational or bio-sampling study is allowed.
  9. Active systemic bacterial, viral, or fungal infection.
  10. Nausea and vomiting ≥ National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0 Grade 2 (for those not controlled by supportive care), malabsorption requiring supplementation, or significant bowel or stomach resection that would preclude adequate absorption of tovorafenib.
  11. Patient has CTCAE v5.0 Grade 3, creatine phosphokinase (CPK) elevation (> 5 × ULN - 10 × ULN).
  12. Patients who are neurologically unstable despite adequate treatment (e.g., uncontrolled seizures).
  13. Pregnancy or lactation.
  14. History of drug reaction with eosinophilia and systemic symptoms (DRESS) syndrome or Stevens Johnsons syndrome (SJS). Patients with hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any other excipient present in the pharmaceutical form of the investigational medicinal product.
  15. Other unspecified reasons that, in the opinion of the investigator, make the patient unsuitable for enrollment.

Ages: 0 Weeks to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2027-03-21 (Estimated); Study Completion 2029-03-21 (Estimated)

PRIMARY OUTCOMES:
MTD/RP2D | 2 years
  To determine the maximum tolerated dose (MTD/RP2D) of combination of vinblastine + tovorafenib for children with recurrent/progressive LGGs.
Safety and Tolerability | 2 years
  To assess safety and tolerability of combination of vinblastine and tovorafenib in pediatric patients with recurrent/progressive LGG through documentation of number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Overall response rate | 2 years
  To determine overall response rate (ORR) of CR, PR and MR in patients with LGG treated with combination of vinblastine + tovorafenib by RANO-LGG criteria.

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax vinblastine and tovorafenib) | 5 years (to complete analyses)
  To characterize pharmacokinetics of tovorafenib and vinblastine in combination in the study population. The following PK parameters will be determined for each agent: Cmax, Tmax, AUC and reported using descriptive summary statistics
Pharmacokinetics (AUC of vinblastine and tovorafenib) | 5 years (to complete analyses)
  To characterize pharmacokinetics of tovorafenib and vinblastine in combination in the study population. The following PK parameters will be determined for each agent: Cmax, Tmax, AUC and reported using descriptive summary statistics
Progression free survival | 3-year
Duration of response | 3 years
  DOR for patients with CR, PR or MR based on RANO-LGG criteria
Clinical Benefit rate | 3 years
  CR, PR and MR plus stable disease which lasts a minimum of 24 weeks by RANO-LGG criteria

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Morgenstern, Study Director — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada